CLINICAL TRIAL: NCT02818140
Title: Ultrasound-guided Transmuscular Quadratus Lumborum Block for Elective Percutaneous Nephrolithotomy
Brief Title: Ultrasound-guided Transmuscular Quadratus Lumborum Block for Percutaneous Nephrolithotomy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Zealand University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2015-004770-16
Record Dates: First submitted 2016-06-27; First posted 2016-06-29 (Estimated); Last update posted 2018-03-22 (Actual); Status verified 2018-03

CONDITIONS: Kidney Stone
Keywords: Postoperative pain; Transmuscular quadratus lumborum block; Block; Ropivacaine; TQL; percutaneous nephrolithotomy; PNL; Ultrasound-guided
MeSH Terms: conditions — Kidney Calculi; Pain, Postoperative; Bites and Stings | interventions — Ropivacaine; Sodium Chloride; Ultrasonography

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ropivacaine TQL block (Active Comparator): Unilateral single shot ultrasound-guided TQL block with 30 ml of ropivacaine 0.75%
  Interventions: Procedure: Ropivacaine TQL block; Drug: Ropivacaine; Device: Ultrasound
- Placebo TQL block (Placebo Comparator): Unilateral single shot ultrasound-guided TQL block with 30 ml saline 0.9%
  Interventions: Procedure: Saline TQL block; Drug: Saline; Device: Ultrasound

INTERVENTIONS:
Procedure: Ropivacaine TQL block — Unilateral ultrasound-guided TQL block with 30 mL ropivacaine 0.75% 30 min prior to the surgical procedure
  Other Names: Naropin
  Arms: Ropivacaine TQL block
Procedure: Saline TQL block — Unilateral ultrasound-guided TQL block with 30 mL of saline 0,9% 30 min prior to the surgical procedure
  Arms: Placebo TQL block
Drug: Ropivacaine
  Arms: Ropivacaine TQL block
Drug: Saline
  Arms: Placebo TQL block
Device: Ultrasound

SUMMARY:
Patients undergoing percutaneous nephrolithotomy (PNL) suffer from acute postoperative pain, despite a multimodal analgesic regime.

We hypothesize that active (ropivacaine) transmuscular quadratus lumborum (TQL) block will significantly reduce postoperative opioid consumption and pain following PNL operation compared with placebo (saline) TQL block.

The aim of this study is to investigate the effect of ultrasound-guided (USG) TQL block concurrent with a multimodal analgesic regime compared to the multimodal analgesic regime alone (and placebo TQL block) in a randomized and placebo controlled design.

DETAILED DESCRIPTION:
Patients undergoing percutaneous nephrolithotomy (PNL) suffer from acute postoperative pain, despite a multimodal analgesic regime, and the patients receive considerable amounts of long lasting opioids. For the patients this greatly increase the risk of experiencing the adverse effects of opioids.

The ultrasound-guided (USG) transmuscular quadratus lumborum (TQL) block is a single dosage of local anesthetic (LA) delivered in the plane between the psoas major muscle and the quadratus lumborum muscle. LA spreads cephalad into the thoracic paravertebral space to reach the somatic ventral rami (intercostal nerves) and the thoracic sympathetic trunk. The TQL block can reduce visceral pain and pain originating from the abdominal wall and has an expected duration of analgesic efficacy of 24 hours.

The aim of this study is to investigate the efficacy of the active USG TQL block together with the multimodal analgesic regime to reduce postoperative opioid consumption and pain compared to placebo USG TQL block and the multimodal analgesic regime in a randomized and placebo controlled design.

ELIGIBILITY:
Inclusion Criteria:

Scheduled for elective PNL operation in general anaesthesia with propofol and remifentanil.

Received oral and written information about the trial Signed the informed consent American Society of Anesthesiologists (ASA) classification 1-3

Exclusion Criteria:

Cannot cooperate Does not speak or understand Danish Allergy towards drugs used in the trial Large daily consumption of opioids Known alcohol or drug abuse Difficulty or inability to visualize the relevant muscular or fascial structures necessary to perform the USG-TQL block Pregnancy

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-07; Primary Completion 2018-03 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Total morphine consumption | 6 hours postoperatively
  Morphine consumption in the first 6 hours postoperatively - data from PCA pump and patient medical record

SECONDARY OUTCOMES:
Total morphine consumption | 15 min, 30 min, 1 h, 2h, 4h, 6h, 12h, 18h, 24 hours postoperatively
  Data from PCA pump and patient electronic file
Pain score at rest (NRS 0-10/10) | 15 min, 30 min, 1 h, 2h, 4h, 6h, 12h, 18h, 24 hours postoperatively
  Pain score NRS
Pain score at sitting position (NRS 0-10/10) | 15 min, 30 min, 1 h, 2h, 4h, 6h, 12h, 18h, 24 hours postoperatively
  Pain score NRS
Time to first ambulation - get out of bed | 0-24 hours postoperatively
  Time to first ambulation from bed to walk on the floor
Opioid side effects (nausea, vomiting) | 0-24 hours postoperatively
  PONV, number of episodes, antiemetics
NRS score during application of the TQL block (NRS 0-10/10) | intraoperative
  Procedure discomfort

CONTACTS AND LOCATIONS:
Overall Officials: Mette Dam, MD, PhD Fellow, Principal Investigator — Zealand University Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hansen CK, Dam M, Bendtsen TF, Borglum J. Ultrasound-Guided Quadratus Lumborum Blocks: Definition of the Clinical Relevant Endpoint of Injection and the Safest Approach. A A Case Rep. 2016 Jan 15;6(2):39. doi: 10.1213/XAA.0000000000000270. No abstract available. PMID 26771297
- [Background] Dam M, Hansen CK, Borglum J, Chan V, Bendtsen TF. A transverse oblique approach to the transmuscular Quadratus Lumborum block. Anaesthesia. 2016 May;71(5):603-4. doi: 10.1111/anae.13453. No abstract available. PMID 27072772
- [Derived] Dam M, Hansen CK, Poulsen TD, Azawi NH, Wolmarans M, Chan V, Laier GH, Bendtsen TF, Borglum J. Transmuscular quadratus lumborum block for percutaneous nephrolithotomy reduces opioid consumption and speeds ambulation and discharge from hospital: a single centre randomised controlled trial. Br J Anaesth. 2019 Aug;123(2):e350-e358. doi: 10.1016/j.bja.2019.04.054. Epub 2019 May 30. PMID 31153628